CLINICAL TRIAL: NCT05564533
Title: Neurophysiological Effects of Interoceptive Compassion Training
Brief Title: Heart-Smile Training Intensive Introduction Program
Acronym: HST-IIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other); Korea Advanced Institute of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHA-IRB-21-22-100
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart-Smile Training Intensive Introductory Program (HST-IIP) Group (Experimental): The HST-IIP group will complete the Heart-Smile Training Intensive Introductory Program during weeks 1 through 4 of the study.
  Interventions: Behavioral: Heart-Smile Training Intensive Introduction Program (HST-IIP)
- Waitlist Control Group (No Intervention): The waitlist arm will not complete any intervention during their time in the study. They will continue their treatment as usual without any change in their therapy session or medication. After their post study visits are complete, they will have the opportunity to participate in Mindfulness-Based Intervention courses through the Cambridge Health Alliance Center for Mindfulness and Compassion.

INTERVENTIONS:
Behavioral: Heart-Smile Training Intensive Introduction Program (HST-IIP) — Heart-Smile Training (HST) is an interoceptive compassion program designed to develop the qualities of compassion, empathy, and kindness for oneself and others with a focus on interoceptive awareness. It is unique from other compassion trainings in its focus on 1) embodiment of warmth and tenderness of compassionate feeling with a compassionate body scan meditation, 2) development of an "authentic presence," characterized by a warm feeling of loosened attachment to ego-based self, and 3) cultivation of joy triggered by genuine smile to oneself. HST-IIP is a 3-day/4-week/1-day interoceptive compassion program that shares the same core elements and practices as HST 3-day intensive program. Unlike HST, the format of the HST-IIP has an extended duration to develop self-regulation through the cultivation of emotional and behavioral regulation.
  Arms: Heart-Smile Training Intensive Introductory Program (HST-IIP) Group

SUMMARY:
Heart-Smile Training (HST) is a compassion and loving-kindness-based intensive introduction program consisting of a 3-day retreat, 4-weeks of weekly 2 hour meetings, and a 1-day final retreat. This study is a randomized controlled trial study to evaluate the effectiveness of Heart-Smile Training as compared to the passive control group on measures of neural, physiological, and clinically-relevant outcomes among individuals with symptoms of depression. Participants will be randomized to either the HST group or a waitlist control group. Both groups will complete assessments before and after HST including electroencephalography (EEG), electrocardiogram (EKG), electrodermal activity tests, and self-report surveys. All study activities except surveys will be conducted in person.

DETAILED DESCRIPTION:
This will be a randomized controlled trial with two arms: Heart-Smile Training Intensive Introduction Program (HST-IIP) vs. a waitlist control group. These two arms will be compared on measures of neural, physiological, and clinically-relevant outcomes.

The investigators will enroll up to 50 adult volunteers from the general population from the ages of 18 to 65 with depression, with Computerized Adaptive Test- Depression Inventory (CAT-DI) scores from 35-75. Volunteers interested in the study will be consented and screened for their eligibility. Eligible participants will be randomized to join either the HST-IIP arm or a waitlist control arm after completing all baseline assessments and the EEG session.

Both the HST-IIP and waitlist arm will complete a baseline measurement session between study weeks -3 to 0, before starting any group sessions. Prior to completing the baseline measurement section, they will be randomized to either HST-IIP or the waitlist arm. Participants enrolled in the HST-IIP arm will join the intervention group between week 1 to 5. The waitlist arm will not join any program between week 1 to 5. They will continue their treatment as usual without any change in their therapy session or medication. Both arms will complete weekly survey measures for 5 weeks. Both arms will then complete a post measurement session during study weeks 5 to 7.

At both baseline and post-intervention measurement sessions, all participants will complete in-person study tasks and remote surveys. In-person study visits will include neurophysiological measures; EEG, EKG, skin conductance, and respiration rate measures and will take place at the Spaulding Rehabilitation Hospital/Mass General Brigham in Charlestown, MA. Remote self-report surveys will be completed by participants during baseline and post-measurement either at home through a link secure to the Cambridge Health Alliance (CHA) REDCap database sent via email or using an electronic device at the CHA Center for Mindfulness and Compassion.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient English fluency to understand procedures and questionnaires
* Ability to provide informed consent
* Mild to moderately severe depression (CAT-DI score 35-75) (Achtyes et al., 2015; Gibbons et al., 2012)

Exclusion Criteria:

* Cognitive inability as demonstrated by Montreal Cognitive Assessment (MOCA) <24 OR the inability to complete consent quiz and baseline assessments (Nasreddine et al., 2005);
* Current participation in another research study;
* Unavailable or unable to participate in planned dates for the HST-IIP sessions;
* Expected hospitalization during the study period, including second and third trimester pregnancy at screening;
* Expected incarceration during the study period;
* Previous experience with mindfulness or other mind-body practices, defined as more than 10 minutes of practice per day, more than 5 days a week for the past 6 months; participation in an 8-week mindfulness group program in the last 2 years; or participation in a meditation retreat longer than 1 day in the past 2 years;
* Inability to successfully complete in-person study sessions with EEG, EKG, respiration rate, and skin conductance response measurement as determined by the principal investigator;
* Inability to participate safely in the study intervention and without disrupting the group (in the opinion of principal investigator OR meeting any of the following criteria):
* Active psychosis defined by a PSY-S-CAT score > 60 (from the CAT-MH assessment) will trigger the requirement of a clinical assessment prior to participation in the program (Achtyes et al., 2015)
* Bipolar I disorder history or severe level of mania on CAT-MH (score >70) (Achtyes et al., 2015): In addition, current use of mood stabilizing medication for bipolar disorder.
* Severe depression, indicated by CAT-DI > 75 (Achtyes et al., 2015; Gibbons et al., 2012)
* Acute homicidality with plan and/or intent;
* Acute suicidality or hospitalization for suicide attempt or self-harm within three months of the enrollment period;
* Severe Borderline Personality Disorder or other severe personality disorder that may lead to disruptions within the group; and/or
* Moderate or severe Substance Use Disorder. In addition, reported use of illicit drugs (i.e., cocaine, methamphetamine) OR non-prescribed controlled medications (opioids, stimulants, or benzodiazepines) in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline heartbeat evoked potential (HEP) at 5 weeks | Up to 11 weeks
  HEP has been used as a marker to assess interoceptive awareness between depressed individuals and normal control (MacKinnon et al., 2013). The second primary outcome is to evaluate the effects of HST-IIP on EEG heartbeat evoked potentials (HEP) and the correlation between the pre- versus post-intervention changes in HEP amplitude and changes in depression severity.

SECONDARY OUTCOMES:
Change from Baseline Gamma Band Frequency at 5 weeks | Up to 11 weeks
  Gamma band frequency (>35 Hz) has been demonstrated as an objective measure of meditation experience across techniques (Braboszcz et al., 2017) and is associated with positive emotionality and enhanced affective regulation. Therefore, the primary outcome measure is an EEG measure of amplitude (power) in the gamma frequency band (>35 Hz), during both resting and compassionate state induction, from baseline to post-intervention.
Change from Baseline Depression (CAT-DI) at 5 weeks | Up to 11 weeks
  Computerized Adaptive Test-Depression Inventory (CAT-DI) will be used to assess the depression severity (Achtyes et al., 2015; Gibbons et al., 2012).
Change from Baseline High Frequency Heart Rate Variability (HF-HRV) at 5 weeks. | Up to 11 weeks
  HRV is an autonomic biomarker of cardiovagal modulation. HRV will be calculated from EKG which will be recorded with EEG co-synchronously.

OTHER OUTCOMES:
Change from Baseline Skin Conductance Response at 5 weeks | Up to 11 weeks
  Skin conductance is a psychophysiological measure of sympathetic nervous system activity. Skin conductance response (SCR) will be measured with EEG co-synchronously.
Change from Baseline Clinically Relevant Psychological Data at 5 weeks | Up to 11 weeks
  Clinically Relevant Psychological outcome measures include assessments of mindfulness, self-compassion, interoceptive awareness, interoceptive appreciation, difficulties in emotional regulation, quality of life, gratitude, anxiety, depression, stress, purpose in life, and social connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance Center for Mindfulness and Compassion
Locations (1):
- Cambridge Health Alliance Center for Mindfulness and Compassion, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achtyes ED, Halstead S, Smart L, Moore T, Frank E, Kupfer DJ, Gibbons R. Validation of Computerized Adaptive Testing in an Outpatient Nonacademic Setting: The VOCATIONS Trial. Psychiatr Serv. 2015 Oct;66(10):1091-6. doi: 10.1176/appi.ps.201400390. Epub 2015 Jun 1. PMID 26030317
- [Background] Braboszcz C, Cahn BR, Levy J, Fernandez M, Delorme A. Increased Gamma Brainwave Amplitude Compared to Control in Three Different Meditation Traditions. PLoS One. 2017 Jan 24;12(1):e0170647. doi: 10.1371/journal.pone.0170647. eCollection 2017. PMID 28118405
- [Background] Gibbons RD, Weiss DJ, Pilkonis PA, Frank E, Moore T, Kim JB, Kupfer DJ. Development of a computerized adaptive test for depression. Arch Gen Psychiatry. 2012 Nov;69(11):1104-12. doi: 10.1001/archgenpsychiatry.2012.14. PMID 23117634
- [Background] MacKinnon S, Gevirtz R, McCraty R, Brown M. Utilizing heartbeat evoked potentials to identify cardiac regulation of vagal afferents during emotion and resonant breathing. Appl Psychophysiol Biofeedback. 2013 Dec;38(4):241-55. doi: 10.1007/s10484-013-9226-5. PMID 23824262
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Derived] Kim E, Joss D, Marin F, Anzolin A, Gawande R, Comeau A, Ellis S, Bumpus C, Cahn BR, Kim MWD, Napadow V, Schuman-Olivier Z. Protocol for a Pilot Study on the Neurocardiac Mechanism of an Interoceptive Compassion-Based Heart-Smile Training for Depression. Glob Adv Integr Med Health. 2024 Nov 3;13:27536130241299389. doi: 10.1177/27536130241299389. eCollection 2024 Jan-Dec. PMID 39498312